CLINICAL TRIAL: NCT04205019
Title: A 3 Months Open Phase I Study to Assess the Safety of the Intrathecal Application of Neuro-Cells in End Stage (Chronic) Traumatic Spinal Cord Injury Patients
Brief Title: Safety Stem Cells in Spinal Cord Injury
Acronym: SSCiSCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuroplast (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2019SCI04
Record Dates: First submitted 2019-11-21; First posted 2019-12-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-03

CONDITIONS: Spinal Cord Injuries
Keywords: Traumatic Spinal Cord Injury; Stem Cells
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: TSCI patients are treated once at start of the study and followed up for 3 months to characterize and confirm safety of intrathecal administration of Neuro-Cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuro-Cell group (Experimental): Patient receives treatment once at start of study and followed up for safety.
  Interventions: Biological: Neuro-Cells

INTERVENTIONS:
Biological: Neuro-Cells — Neuro-Cells is an autologous fresh stem cells containing product which modulates the secondary inflammation following a TSCI, reduces apoptosis (cell death) in the injured spinal cord, reduces scar tissue formation in the damaged spinal cord and creates a cell regenerative environment in the injured spinal cord.

SUMMARY:
Mono-center, open label study to investigate the safety of Neuro-Cells in 10 end stage (chronic) traumatic spinal cord injury (TSCI) patients, when administered once intrathecally. TSCI is a rare disease without cure perspectives and Neuro-Cells is an autologous fresh stem cells containing product (one batch / one patient).

DETAILED DESCRIPTION:
This phase I clinical study is an open clinical trial to investigate the safety of the intrathecal application of Neuro-Cells in the treatment of end stage (chronic), traumatic complete (AIS grade A) and incomplete (AIS grade B/C) SCI patients. To that purpose, after inclusion in this study >1 year and less than 5 years after their SCI-event, 10 patients will be included. All patients are invited to visit the trial hospital every month during this 3-months study for appreciation of their possible (S)AEs and/or SUSARs, for physical examination and a biochemical analysis of their blood/urine. Day 0 and day 90 they also undergo a comprehensive neurological examination, the AISIAms, ASIAss and Pain perception.

Finally, the participants are also invited to undergo neurological examinations at day 360 and 720. The purpose of this neurological assessment is to explore in patients if a late administration of Neuro-Cells may have some beneficial effects on the neurological condition of the chronic SCI patient.

All patients undergo a BM harvesting at the start of their participation in the study and will undergo one LP, performed to administer Neuro-Cells. The study is open and descriptive, and no randomization takes place. All patients are followed up until approximately 3 months after the time of administration. After these 3 months, the safety part of this study ends. Patients are invited for a neurological assessment 9 months later (day 360) to explore if Neuro-Cells may have a beneficial effect when given to end stage patients with a traumatic SCI.

The safety part of the study is completed when the last patient finishes his/her visit at day 90. The explorative part of the study ends approximately one year after the time of inclusion at day 720.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 - 40 years
2. Complete (AIS grade A) or incomplete (AIS grade B) TSCI (ISNCSCI-assessed) at time of recruitment
3. Level of injury between C5 to T12
4. Voluntary signed informed consent by patients and Investigator before any trial-related procedures are performed

Exclusion Criteria:

1. SCI AIS grade D or E at the start of enrolment
2. Allergic to mice antibodies and/or iron-dextran
3. Level of SCI above C5 or below T12
4. Positive HIV, hepatitis B or C serology
5. Positive Lues test
6. Total Nuclear Cell (TNC) count < 1x109 TNC
7. Cancer, brain injury, disturbed consciousness, signs/symptoms of neurodegenerative disorder (e.g. stroke, amyotrophic lateral sclerosis, multiple sclerosis etc), diabetes mellitus type 1, renal or cardiac insufficiency based on anamnesis history and at the investigator's discretion
8. Any concomitant treatment or medication that interferes with the conduct of the trial, such as immune-suppressive medication or other medication (especially methotrexate, cyclosporine, and corticosteroids have to be avoided) known to interact with the anti-inflammatory and immune-modulative actions of stem cells (non-steroid anti-inflammatory drugs (NSAIDs) are allowed)
9. Abuse of alcohol (daily consumption of more than 2 units of alcohol containing drinks) or illicit drugs (e.g. heroin, cocaine, XTC)
10. Individuals that belong to vulnerable population groups
11. Females with childbearing potential without using adequate birth control methods (e.g. contraceptive pills, intrauterine devices (IUD), contraceptive injections (prolonged-release), subdermal implantation, vaginal ring or transdermal patches), and/or being pregnant or in the lactation period
12. Participation in any clinical trial (with exemption of descriptive studies with questionnaires and no active intervention) within the previous 30 days before enrolment, or simultaneous participation in such trial
13. Patients with extreme comorbidity before or after the TSCI are excluded at discretion of the PI
14. Patients who are unable to comply with the requirements of this clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Characterize and confirm safety of intrathecal administration of Neuro-Cells by ISNCSCI checklist | 3 months
  checklist in which the physician focusses on the spinal cord
Characterize and confirm safety of intrathecal administration of Neuro-Cells assessed by blood | 3 months
  Measuring biochemical blood variables
Characterize and confirm safety of intrathecal administration of Neuro-Cells assessed by urine | 3 months
  Measuring biochemical urine variables
Characterize and confirm safety of intrathecal administration of Neuro-Cells by adverse events | 3 months
  Severity of adverse events (if applicable)

SECONDARY OUTCOMES:
The effect of late administration of Neuro-Cells by change in American Spinal Injury Association motor scale score | 24 months
  Change in the ASIAms score from baseline at 3 months, 12 months and 24 months. Higher score means more change.
The effect of late administration of Neuro-Cells by change in American Spinal Injury Association sensory scale score | 24 months
  Change in the ASIAss from baseline at 3 months, 12 months and 24 months. Higher score means more change.
Investigate the effect of Neuro-Cells on the autonomic neurological dysfunction | 24 months
  International Standards for Neurological Classification of Spinal Cord Injury assessment , a higher score means improvement
The effect of Neuro-Cells on the sensory neurological dysfunction | 24 months
  International Standards for Neurological Classification of Spinal Cord Injury assessment , a higher score means improvement
The effect of Neuro-Cells on the daily activity level as measured by the Pain basic data set | 24 months
  Pain basic data set using scale with the higher the mesaure the more pain, assessed by physician.
The effect of Neuro-Cells on change in pain assessed by the pain basic data set scale. | 24 months
  Pain basic data set using scale with the higher the mesaure the more pain, assessed by physician.
The effect of Neuro-Cells on pain-reducing medication by looking at change in prescribed medication | 24 months
  Documentation of concomitant medication and the change in prescriptions. Lower dose, less medication is bigger effect.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes P de Munter, MSc, Study Director — CEO Neuroplast
Locations (1):
- Hospital Nacional de Parapléjicos, Toledo, Castille-La Mancha, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuroplast Press Release Primary Safety Results — https://062a517c-8890-4012-ae04-9f771a08c58d.filesusr.com/ugd/6064f5_f22feb9cc2d9412596823d092a3b119c.pdf